CLINICAL TRIAL: NCT04809298
Title: Prospective, Randomized, Controlled, Parallel Group Study to Compare a New Needle Navigation Device for CT-guided Interventions to the Conventional Free-hand Method
Brief Title: Comparison of a New Needle Navigation Device for CT-guided Interventions to the Conventional Free-hand Method
Acronym: PunctureCube
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Luca Remonda (Other)
Responsible Party: Sponsor-Investigator, Luca Remonda, Prof. Dr. med., Kantonsspital Aarau
Organization: Kantonsspital Aarau (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Puncture Cube
Record Dates: First submitted 2021-03-05; First posted 2021-03-22 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Lumbar Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, controlled, parallel group study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Free-hand lumbar punction (Other): Diagnostic or therapeutic CT-guided intervention for lumbar pain management using the free-hand method.
  Interventions: Device: Free-hand therapeutic CT-guided punction for lumbar pain
- Puncture Cube (Active Comparator): Diagnostic or therapeutic CT-guided intervention for lumbar pain management using the Puncture Cube® as a needle navigation device.
  Interventions: Device: Puncture Cube

INTERVENTIONS:
Device: Free-hand therapeutic CT-guided punction for lumbar pain — Diagnostic or therapeutic CT-guided intervention for lumbar pain management using the Puncture Cube® as a needle navigation device.
  Arms: Free-hand lumbar punction
Device: Puncture Cube — Diagnostic or therapeutic CT-guided intervention for lumbar pain management using the Puncture Cube® as a needle navigation device.
  Arms: Puncture Cube

SUMMARY:
In a prospective, randomized, controlled, parallel group study the accuracy, intervention time and radiation dose of CT-guided punctures using the Puncture Cube® will be compared to the conventional free-hand method in patients requiring a percutaneous diagnostic or therapeutic CT-guided intervention for lumbar pain (facet joint-, nerve root-, epidural infiltrations at the lumbar/lumbosacral level).

DETAILED DESCRIPTION:
Computed tomography (CT)-guided interventions for diagnostic and therapeutic purposes are standard approaches in clinical routine (e.g. in patients with low back pain). Numerous CT needle navigation systems have been developed with the aim to improve accuracy (and thus safety) of punctures while decreasing radiation exposure and procedure time. Their usability in clinical routine is limited either because of high sensitivity to interference, high expenses, bulkiness, or incompatibly with daily clinical practice and thus increasing procedure time and workflow complexity. The Puncture Cube® takes into account all these requirements. Furthermore, in an in vitro-phantom study (study submitted for publication), punctures with the Cube were found to be faster and more accurate compared to the free-hand conventional method.

In a prospective, randomized, controlled, parallel group study the accuracy, intervention time and radiation dose of CT-guided punctures using the Puncture Cube® will be compared to the conventional free-hand method in patients requiring a percutaneous diagnostic or therapeutic CT-guided intervention for lumbar pain (facet joint-, nerve root-, epidural infiltrations at the lumbar/lumbosacral level).

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring a percutaneous therapeutic CT-guided intervention for
* lumbar pain (joint-, nerve root-, epidural infiltrations at the lumbar/lumbosacral level)
* age ≥ 18 years
* Signed informed consent prior to intervention

Exclusion Criteria:

* Patients suffering from severe obesity (BMI > 30 kg/m2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Puncture accuracy | during procedure time approximately 30 min.
  Assessment of puncture accuracy (distance and angle error between planned and achieved trajectory)

SECONDARY OUTCOMES:
Number of control acquisitions to achieve target | during procedure time approximately 30 min.
  Number of control acquisitions to achieve target
Assessment of radiation dose | during procedure time approximately 30 min.
  Assessment of radiation dose
Assessment of intervention time | during procedure time approximately 30 min.
  Assessment of intervention time

CONTACTS AND LOCATIONS:
Overall Officials: Luca Remonda, Prof., Principal Investigator — Department of Neuroradiology, Kantonsspital Aarau
Locations (1):
- Department of Neuroradiology, Kantonsspital Aarau, Aarau, Canton of Aargau, Switzerland

IPD SHARING:
Plan to Share IPD: No